CLINICAL TRIAL: NCT04606069
Title: Clinical Trial on the Safety and Efficacy of Regadenoson for Moderate to Severe COVID-19 Adult Patients
Brief Title: Treat COVID-19 Patients With Regadenoson
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Christine Lau, Dr. Robert W. Buxton Professor and Chair Department of Surgery, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HP-00091372
Record Dates: First submitted 2020-10-26; First posted 2020-10-28 (Actual); Results first posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-02

CONDITIONS: COVID-19; Lung Inflammation
MeSH Terms: conditions — COVID-19; Pneumonia | interventions — regadenoson; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Arm (Experimental): Regadenoson will be given intravenously as 5 ug/kg loading dose (up to 400 mg/patient) over 30 mins (to avoid unpleasant side effects sometimes associated with the rapid bolus injection of Regadenoson), followed by a continuous slow infusion (1.44micrograms/kg/hour) with the use of a pediatric infusion pump for 6 hours.
  Interventions: Drug: Regadenoson
- Control Arm (Placebo Comparator): The same volume of saline will be given intravenously for 30 mins followed by a continuous infusion for 6 hours.
  Interventions: Other: Placebo Control

INTERVENTIONS:
Drug: Regadenoson — Regadenoson will be given intravenously as 5 ug/kg (up to 400 mg/patient) loading dose over 30 mins (to avoid unpleasant side effects sometimes associated with the rapid bolus injection of Regadenoson), followed by a continuous slow infusion (1.44micrograms/kg/hour) with the use of a pediatric infusion pump for 6 hours.
  Other Names: LEXISCAN,
  Arms: Active Arm
Other: Placebo Control — The same volume of saline will be given intravenously for 6 and half hours.
  Other Names: Saline
  Arms: Control Arm

SUMMARY:
More than 17 million people have been infected and more than 677K lives have been lost since the COVID-19 pandemic. Unfortunately, there is neither an effective treatment nor is there a vaccination for this deadly virus. The moderate to severe COVID-19 patients suffer acute lung injury and need oxygen therapy, and even ventilators, to help them breathe. When a person gets a viral infection, certain body cells (inflammatory/immune cells) get activated and release a wide range of small molecules, also known as cytokines, to help combat the virus. But it is possible for the body to overreact to the virus and release an overabundance of cytokines, forming what is known as a "cytokine storm". When a cytokine storm is formed, these cytokines cause more damage to their own cells than to the invading COVID-19 that they're trying to fight. Recently, doctors and research scientists are becoming increasingly convinced that, in some cases, this is likely what is happening in the moderate to severe COVID-19 patients. The cytokine storm may be contributing to respiratory failure, which is the leading cause of mortality for severe COVID-19 patients. Therefore, being able to control the formation of cytokine storms will also help alleviate the symptoms and aid in the recovery of severe COVID-19 patients.

DETAILED DESCRIPTION:
The investigators reason that Regadenoson treatment will reduce COVID-19-induced lung injury by inhibiting hyperinflammation. Our overarching goal is to demonstrate that Regadenoson treatment increases survival by reducing hyperinflammation and pulmonary function. The investigators will test the hypothesis that Regadenoson elicits clinical improvement and enhances survival compared to placebo control patients with COVID-19. The investigators hypothesize that the survival benefit of Regadenoson will be additive or synergistic with the anti-viral drug, Remdesivir. Remdesivir and Dexamethasone are currently standard of care and would remain so.

Specific Aim 1: will determine the initial high dose followed by low dose continuous infusion that is safe and feasible in moderate to severe COVID-19 patients. Even if the dosages that the investigators will use in moderate to severe COVID-19 patients has been proved to be safe in myocardial perfusion imaging patients, sickle cells disease and lung transplantation patients, it is still unclear whether it is safe in COVID-19 patients. Therefore, our primary endpoint for this Aim will be safety. For the first 6 patients, the investigators will be looking at any drug related side effects and toxicity of Regadenoson as the investigators did in lung transplantation trial.

Specific Aim 2: will determine the potential efficacy of Regadenoson infusion in moderate to severe COVID-19 patients. If Regadenoson infusion is safe and feasible in the moderate to severe COVID-19 patients in Aim 1, the investigators will test its efficacy in 34 moderate to severe COVID-19 patients in a randomized controlled trial of regadenoson versus placebo control. The primary endpoints of this specific aim are: 1) Proportion of patients alive and free of respiratory failure through the 30 day trial. Respiratory failure is defined based on resource utilization requiring at least 1 of the following modalities, 2) Endotracheal intubation and mechanical ventilation, 3) Oxygen delivered by high-flow nasal cannula (heated, humidified, oxygen delivered via reinforced nasal cannula at flow rates >20L/min with fraction of delivered oxygen ≥0.5), 4) Noninvasive positive pressure ventilation or CPAP, 5) ECMO.

Specific Aim 3: will explore the mechanisms of the effects of Regadenoson infusion in moderate to severe COVID-19 patients. If Regadenoson is proved to be effective on treating moderate to severe COVID-19 patients in Aim 2, the investigators will continue the study in this Aim. The investigators will measure 1) the plasma levels of Regadenoson in the collected blood samples (these will be done only on the first 6 patients as the investigators need specific time points and want to limit non routine blood draws); 2) the levels of pro-inflammatory cytokines (TNF-α, IL-1, IL-6, IL-12, IL-8, INF-γ, etc) and anti-inflammatory cytokines ( IL-4 and IL-10), and 3) the levels of matrix metalloproteinase-9 (MM-9) and tissue inhibitor of metalloproteinase-1 (TIMP-1) in blood samples which will be collected from COVID-19 patients at prior baseline lab draws and also next day am routine labs. For the first 6-patients the investigators will ask for 2- additional study lab draws, one at the conclusion of the 30-min infusion and one at 4-hours into the 6-hours slow continuous infusion. The investigators may limit this to 3 if there are no dose limiting toxicities. The investigators are asking for up to 6 in the safety aim 1 in case one of the 3 has a dose limiting toxicity the investigators would then provide to 6 total. 5 of 6 would need to be without dose limiting toxicity to continue with the additional 34 patients.

ELIGIBILITY:
Inclusion Criteria:

* Age: adults 18 years and older
* Laboratory-confirmed COVID-19+ by RT-PCR
* Moderate to Severe COVID-19 patients according to FDA's COVID-19 treatment guideline on Management of Persons with COVID-19: Moderate illness is defined as individuals who have evidence of lower respiratory disease by clinical assessment or imaging and a saturation of oxygen (SpO2) >93% on room air at sea level. Severe Illness is defined as individuals who have respiratory frequency >30 breaths per minute, SpO2 ≤ 93% on room air at sea level, ratio of arterial partial pressure of oxygen to fraction of inspired oxygen (PaO2/FiO2) <300, or lung infiltrates >50%
* Written informed consent must be obtained before any study procedure is performed.

Exclusion Criteria:

* Pregnant or breastfeeding women
* Symptoms or signs of acute myocardial ischemia
* Sinoatrial (SA) and Atrioventricular (AV) Nodal Block/dysfunction
* Symptoms or signs of Atrial Fibrillation/Atrial Flutter
* History of Hypotension
* History of severe hypertension not adequately controlled with anti-hypertensive medications (Systolic blood pressure ≥ 200 mmHg and/or Diastolic blood pressure ≥ 110 mmHg)
* Severe renal impairment defined as glomerular filtration rate (GFR) < 30 ml/min
* History of clinically overt stroke within the past 3 years
* History of seizure disorder
* Pre-existing asthma or chronic obstructive pulmonary disease
* Chronic anti-coagulation or anti-platelet therapy that would preclude surgery (prophylactic aspirin is acceptable)
* 12.Treatment within 30 days with Hydroxychloroquine (HCQ) or Azithromycin
* Treatment with Janus Kinase inhibitors
* Treatment with theophylline or aminophylline within 12 hours of study dosing
* Treatment with Persantine and/or Aggrenox within 5 days
* Other clinical conditions that in the opinion of the investigator would make the subject unsuitable for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine L Lau, MD, MBA, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lau CL, Beller JP, Boys JA, Zhao Y, Phillips J, Cosner M, Conaway MR, Petroni G, Charles EJ, Mehaffey JH, Mannem HC, Kron IL, Krupnick AS, Linden J. Adenosine A2A receptor agonist (regadenoson) in human lung transplantation. J Heart Lung Transplant. 2020 Jun;39(6):563-570. doi: 10.1016/j.healun.2020.02.003. Epub 2020 Feb 13. PMID 32503727
- [Background] Field JJ, Majerus E, Gordeuk VR, Gowhari M, Hoppe C, Heeney MM, Achebe M, George A, Chu H, Sheehan B, Puligandla M, Neuberg D, Lin G, Linden J, Nathan DG. Randomized phase 2 trial of regadenoson for treatment of acute vaso-occlusive crises in sickle cell disease. Blood Adv. 2017 Aug 28;1(20):1645-1649. doi: 10.1182/bloodadvances.2017009613. eCollection 2017 Sep 12. PMID 29296811
- [Background] Zhao Y, Xiao A, diPierro CG, Carpenter JE, Abdel-Fattah R, Redpath GT, Lopes MB, Hussaini IM. An extensive invasive intracranial human glioblastoma xenograft model: role of high level matrix metalloproteinase 9. Am J Pathol. 2010 Jun;176(6):3032-49. doi: 10.2353/ajpath.2010.090571. Epub 2010 Apr 22. PMID 20413683
- [Background] Zhao Y, Sharma AK, LaPar DJ, Kron IL, Ailawadi G, Liu Y, Jones DR, Laubach VE, Lau CL. Depletion of tissue plasminogen activator attenuates lung ischemia-reperfusion injury via inhibition of neutrophil extravasation. Am J Physiol Lung Cell Mol Physiol. 2011 May;300(5):L718-29. doi: 10.1152/ajplung.00227.2010. Epub 2011 Mar 4. PMID 21378024

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment began in Spring of 2021 at the University of Maryland Medical Center. Study staff screened the medical records of COVID 19 positive patients and reviewed to determine study eligibility. Hospitalized COVID-19 patients were approached according to the unit policy (video chat etc).
Groups:
- Regadenoson: Regadenoson will be given intravenously as 5 ug/kg loading dose (up to 400 mg/patient) over 30 mins (to avoid unpleasant side effects sometimes associated with the rapid bolus injection of Regadenoson), followed by a continuous slow infusion (1.44micrograms/kg/hour) with the use of a pediatric infusion pump for 6 hours.
- Placebo: The same volume of saline will be given intravenously for 30 mins followed by a continuous infusion for 6 hours.
Period: Overall Study
Arm/Group | Regadenoson | Placebo
Started | 5 | 0
Completed | 5 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Following the DSMB recommendations, our site was told to enroll 5 participants in the RA group to assess safety. The enrollment was paused for a safety review of the data from the 5 participants. After a review of the preliminary data, we were approved to resume enrollment per the randomization schema. However, at the time of approval peak COVID rates had declined and despite substantial screening efforts, no eligible participants were enrolled. Therefore, the control arm is zero.
Groups:
- Total: Total of all reporting groups
Arm/Group | Regadenoson | Placebo | Total
Number analyzed (Participants) | 5 | 0 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 0 | 4
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (11.4) |  | 53.2 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 4 |  | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 5 |  | 5
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 |  | 1
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 2 |  | 2
  White | 2 |  | 2
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 |  | 5
BMI [Mean (Standard Deviation); unit: Kg/m^2] | 35.5 (6.8) |  | 35.5 (6.8)
Oxygen Supplementation on Admission [Count of Participants; unit: Participants] — Participants were graded clinically based on their oxygen requirements at the time of admission. Participants were either on 2L oxygen via nasal cannula, 6L of oxygen via nasal cannula, or High Flow Nasal Cannula. This information was collected from the electronic medical record based on their initial presentation.
  Participants
    2L NC | 3 |  | 3
    6L NC | 1 |  | 1
    HFNC | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Alive and Free of Respiratory Failure Through the 30-day Trial.
Description: Respiratory failure is defined based on resource utilization requiring at least 1 of the following modalities:
  1. Endotracheal intubation and mechanical ventilation
  2. Oxygen delivered by high-flow nasal cannula (heated, humidified, oxygen delivered via reinforced nasal cannula at flow rates >20L/min with fraction of delivered oxygen ≥0.5)
  3. Noninvasive positive pressure ventilation or CPAP
  4. Whether patient is on ECMO
Time Frame: 30 Days
Population: as for baseline characteristics
Measure: Number; unit: Percentage of of patients alive and free
Arm/Group | Active Arm | Control Arm
Number analyzed (Participants) | 5 | 0
Percentage of of patients alive and free | 100 |

2. Secondary Outcome: Change of the Levels of the Inflammatory Cytokines Prior, During and Post Drug Infusion.
Description: We will collect blood samples of the Regadenoson and Placebo treated patients at baseline, 30mins into infusion, 4 hours into drug infusion and 24 hours post drug infusion. It may also include the daily blood collected on normal standard care base. The inflammatory cytokines, including IL-1 beta, IL-6, IL-4, IL-8, IL-10, IL-12, IL-17, TNF-α, and IFN-γ will be measured using the Luminex™ 100 Multi-analyte System at The UM SOM Cytokine Core Laboratory. The levels of of cytokines will be measure in picogram/milliliter (pg/ml).
Time Frame: Baseline, 30mins into infusion, 4 hours into drug infusion and 24 hours post drug infusion
Population: Cytokine levels were normalized to baseline just prior to RA infusion.
Measure: Mean (95% Confidence Interval); unit: pg/ml
Arm/Group | Regadenoson | Placebo
Number analyzed (Participants) | 5 | 0
pg/ml
  IL-6 - 30 Minutes | 1.53 [0.69 to 3.37] |
  MCP-1 - 30 Minutes | 1.32 [1.11 to 1.58] |
  IL-8 - 30 Minutes | 0.98 [0.60 to 1.59] |
  IL-10 - 30 Minutes | 1.02 [0.73 to 1.43] |
  IL-12p40 - 30 Minutes | 0.76 [0.57 to 1.01] |
  IL-7 - 30 Minutes | 0.80 [0.45 to 1.42] |
  IP-10 - 30 Minutes | 0.77 [0.56 to 1.04] |
  IFN-G - 30 Minutes | 0.90 [0.59 to 1.38] |
  MIP-1A - 30 Minutes | 0.52 [0.20 to 1.35] |
  IL-12p70 - 30 Minutes | 0.76 [0.53 to 1.10] |
  IL-17 - 30 Minutes | 0.49 [0.19 to 1.22] |
  IL-1B - 30 Minutes | 0.49 [0.21 to 1.15] |
  IL-2 - 30 Minutes | 0.45 [0.18 to 1.13] |
  TNF-A - 30 Minutes | 0.45 [0.20 to 1.03] |
  IL-6 - 4hr | 1.23 [0.55 to 2.71] |
  MCP-1 - 4hr | 1.10 [0.92 to 1.32] |
  IL-8 - 4hr | 0.97 [0.60 to 1.59] |
  IL-10 - 4hr | 0.87 [0.62 to 1.22] |
  IL-12p40 - 4hr | 0.81 [0.61 to 1.07] |
  IL-7 - 4hr | 0.78 [0.44 to 1.38] |
  IP-10 - 4hr | 0.76 [0.56 to 1.03] |
  IFN-G - 4hr | 0.73 [0.48 to 1.12] |
  MIP-1A - 4hr | 0.70 [0.27 to 1.80] |
  IL-12p70 - 4hr | 0.70 [0.49 to 1.01] |
  IL-17 - 4hr | 0.60 [0.24 to 1.51] |
  IL-1B - 4hr | 0.50 [0.22 to 1.17] |
  IL-2 - 4hr | 0.47 [0.19 to 1.18] |
  TNF-A - 4hr | 0.47 [0.21 to 1.07] |
  IL-6 - 24hr | 1.53 [0.69 to 3.37] |
  MCP-1 - 24hr | 1.32 [1.11 to 1.58] |
  IL-8 - 24hr | 0.98 [0.60 to 1.59] |
  IL-10 - 24hr | 1.02 [0.73 to 1.43] |
  IL-12p40 - 24hr | 0.76 [0.57 to 1.01] |
  IL-7 - 24hr | 0.80 [0.45 to 1.42] |
  IP-10 - 24hr | 0.77 [0.56 to 1.04] |
  IFN-G - 24hr | 0.90 [0.59 to 1.38] |
  MIP-1A - 24hr | 0.52 [0.20 to 1.35] |
  IL-12p70 - 24hr | 0.76 [0.53 to 1.10] |
  IL-17 - 24hr | 0.49 [0.19 to 1.22] |
  IL-1B - 24hr | 0.49 [0.21 to 1.15] |
  IL-2 - 24hr | 0.45 [0.18 to 1.13] |
  TNF-A - 24hr | 0.45 [0.20 to 1.03] |

ADVERSE EVENTS:
Time Frame: Study participants were monitored for adverse effects from the time of infusion (D1) through Day 30.
Description: Following the DSMB recommendations, our site was told to enroll 5 participants in the RA group to assess safety. The enrollment was paused for a safety review of the data from the 5 participants. After a review of the preliminary data, we were approved to resume enrollment per the randomization schema. However, at the time of approval peak COVID rates had declined and despite substantial screening efforts, no eligible participants were enrolled. Therefore, the control arm is zero.
Arm/Group | Regadenoson | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/0
Other Adverse Events (participants affected / at risk) | 0/5 | 0/0

LIMITATIONS AND CAVEATS:
This study did not include untreated patient controls or have sufficient power to determine if RA reduced mortality or length of stay in the hospital.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-11): https://cdn.clinicaltrials.gov/large-docs/69/NCT04606069/Prot_SAP_000.pdf